CLINICAL TRIAL: NCT00533533
Title: A Phase I/II Trial of Docetaxel and Oxaliplatin in Patients With Advanced Gastric Cancer
Acronym: DO for AGC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Young Suk Park, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-10-047
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2006-11

CONDITIONS: Gastric Cancer
Keywords: Docetaxel,Oxaliplatin; Phase I/II study; Advanced gastric cancer; First line treatment; Advanced gastric cancer with measurable disease
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel, oxaliplatin — Oxaliplatin will be administered in combination with docetaxel as a first-line chemotherapy in advanced gastric cancer patients. Each cycle is repeated every 3 weeks.
  Docetaxel Oxaliplatin Level 1 60 mg/m2/day 1 100 mg/m2/day 1 Level 2 75 mg/m2/day 1 100 mg/m2/day 1 Level 3 75 mg/m2/day 1 130 mg/m2/day 1

SUMMARY:
Gastric cancer is the most common malignancy in Korea. The prognosis of unresectable gastric cancer has been improved by cytotoxic chemotherapy, but median survival rarely exceeds 1 year. New agents such as taxane, irinotecan and oxaliplatin combined with old agents such as 5-FU with or without leucovorin, doxorubicin, cisplatin showed higher response rates in phase II studies. Docetaxel as a single agents showed response rates of 17-24%, and the combination of docetaxel and cisplatin has shown a response rate of 37-56% and overall survival of 9-10.4 months. Oxaliplatin in combination with 5-FU and leucovorin(FOLFOX-6) showed an objective response rate of 50%, which included a 4% complete response. The preclinical studies, oxaliplatin has shown additive or synergistic cytotoxic properties with fluoropyrimidines, thymidylate synthase inhibitors, topoisomerase I inhibitors, microtubule inhibitors and DNA modifying/alkylating agents. The combination of docetaxel and oxaliplatin has been studied previously in the phase I setting in patients with metastatic breast and non-small cell lung cancer. The combination of docetaxel and oxaliplatin is a feasible and well tolerated regimen. Recommended doses were 75mg/m2 for docetaxel on day 1 and 70mg/m2 for oxaliplatin on day 2 without G-CSF support. The aim of this trial is to determine the dose limiting toxicities, maximum tolerated dose(MTD) and efficacy of oxaliplatin and docetaxel as combination chemotherapy in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
Primary objectives :

To define the dose-limiting toxicity and maximum tolerated dose in phase I study To evaluate the overall response rate in phase II study

Secondary objectives :

1. To evaluate the safety and tolerability of the treatment combination.
2. To estimate overall survival.
3. To estimate the time to progression and the duration of overall response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented gastric adenocarcinoma including adenocarcinoma of the esophagogastric junction
* 18 ≤ age ≤ 70
* ECOG performance status of 0 - 2
* At least one definite measurable lesion(s): ≥ 1 cm on spiral CT scan or ≥ 2 cm in physical examination
* Previously untreated metastatic gastric cancer patients or relapsed gastric cancer patients (patients with recurrence at least 6 months from the date of last administration of adjuvant chemotherapy and/or radiation therapy with 5-FU and/or leucovorin containing regimen will be included in the study)
* Written informed consent
* Minimum life expectancy of 12 weeks
* Adequate liver, renal, bone marrow functions as evidence by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; ASAT and/or ALAT < 3 UNL; serum creatinine ≤ 1.5 ULN

Exclusion Criteria:

* Any other malignancies within the past 5 years except skin basal cell cancer or CIS of cervix
* Serious comorbid diseases
* Pregnancy or lactation
* Previous history of drug allergy to one of the drugs in the study regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To define the dose-limiting toxicity and maximum tolerated dose in phase I study To evaluate the overall response rate in phase II study | Two years

SECONDARY OUTCOMES:
1) To evaluate the safety and tolerability of the treatment combination. 2) To estimate overall survival. 3) To estimate the time to progression and the duration of overall response. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, M.D., Ph.D., Principal Investigator — Samsung Medical Center, Seoul, KOREA
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Sulkes A, Smyth J, Sessa C, Dirix LY, Vermorken JB, Kaye S, Wanders J, Franklin H, LeBail N, Verweij J. Docetaxel (Taxotere) in advanced gastric cancer: results of a phase II clinical trial. EORTC Early Clinical Trials Group. Br J Cancer. 1994 Aug;70(2):380-3. doi: 10.1038/bjc.1994.310. PMID 7914428
- [Result] Roth AD, Maibach R, Martinelli G, Fazio N, Aapro MS, Pagani O, Morant R, Borner MM, Herrmann R, Honegger H, Cavalli F, Alberto P, Castiglione M, Goldhirsch A. Docetaxel (Taxotere)-cisplatin (TC): an effective drug combination in gastric carcinoma. Swiss Group for Clinical Cancer Research (SAKK), and the European Institute of Oncology (EIO). Ann Oncol. 2000 Mar;11(3):301-6. doi: 10.1023/a:1008342013224. PMID 10811496
- [Result] Kouroussis C, Agelaki S, Mavroudis D, Kakolyris S, Androulakis N, Kalbakis K, Souglakos J, Mallas K, Bozionelou V, Pallis A, Adamtziki H, Georgoulias V. A dose escalation study of docetaxel and oxaliplatin combination in patients with metastatic breast and non-small cell lung cancer. Anticancer Res. 2003 Jan-Feb;23(1B):785-91. PMID 12680184
- [Result] Louvet C, Andre T, Tigaud JM, Gamelin E, Douillard JY, Brunet R, Francois E, Jacob JH, Levoir D, Taamma A, Rougier P, Cvitkovic E, de Gramont A. Phase II study of oxaliplatin, fluorouracil, and folinic acid in locally advanced or metastatic gastric cancer patients. J Clin Oncol. 2002 Dec 1;20(23):4543-8. doi: 10.1200/JCO.2002.02.021. PMID 12454110